CLINICAL TRIAL: NCT06562374
Title: Low Frequency Ultrasound for Osteoarthritis Healing and Rehabilitation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended by IRB
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0164
Record Dates: First submitted 2024-07-31; First posted 2024-08-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee; Age Related Osteoporosis; Pain; Knee Joint Contracture
Keywords: Pain; Osteo Arthritis Knee; Knee; Ultrasound; Joint mobility
MeSH Terms: conditions — Osteoporosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Frequency Ultrasound (LFU) Intervention (Experimental): Subjects will be given ultrasound at a frequency of 33 kHz with a program of 1.6 seconds on and 1.6 seconds off for 30 min at either a power level of 4 or 10 Pascals to determine which power level is optimal for osteoarthritis. Follow up visits after two-three days will be used to continue therapy.
  Interventions: Device: Low Frequency Ultrasound Therapy

INTERVENTIONS:
Device: Low Frequency Ultrasound Therapy — The ultrasound will be delivered at a frequency of 33 kHz at power levels of 4-10 Pascals with a program of 1.6 seconds on and 1.6 seconds off. The generators will be encased in epoxy within the Osteoarthritis baths. The intervention will be repeated on every second or third day to allow time for healing

SUMMARY:
The purpose of this study is to determine the safety and effectiveness (how well it works) of a new experimental ultrasound bath device that uses low frequency ultrasound (LFU) that may or may not help healing.

DETAILED DESCRIPTION:
This initial study is a pilot study which is going to test the safety and efficacy of the developed ultrasound intervention for osteoarthritis, initially on osteoarthritis of the knee. This study is a pilot study to evaluate two distinct variables. The first is the safety and efficacy of the device, and the second is the potential impact the device may have on patients as their osteoarthritic joints react to the LFU, using patient-reported outcomes associated with this study. The ultrasound will be delivered at a frequency of 33 kHz at power levels of 4-10 Pascals with a program of 1.6 seconds on and 1.6 seconds off. The generators will be encased in epoxy within the Osteoarthritis baths. The intervention will be repeated on every second or third day to allow time for healing

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent in a manner approved by the IRB and is willing and able to comply with the trial procedures.
2. Adults at least ≥40 years of age at the time of consent.
3. Chronic knee pain within the past 6 months.

Exclusion Criteria:

1. Any other arthritic condition clinically classified under ACR guidelines as different from an Osteoarthritic disorder.
2. Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation.
3. History of replacement surgery, acupuncture therapy on the joint/knee under study within the past 6 months, or systemic corticosteroids within the study period and previous 30 days.
4. Subject's vitals are unstable or not in range for a safe study visit.
5. History of fecal incontinence.
6. Vomiting/Diarrheal illness within the past 7 days or at any time during the study.
7. Any clinically significant rash or formation of rashes or open sores, boils or infected wounds two weeks prior to or during the study.
8. Laboratory evidence of infection or colonization with multidrug resistant pathogens in the past 90 days (eg. vancomycin resistant enterococcus, methicillin-resistant Staphylococcus, Candida auris, extended- spectrum beta lactamase bacteria)
9. History of prior non-compliance or the presence or history of psychiatric conditions (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.
10. Females who are pregnant or lactating.
11. Inability to comply with study protocol.
12. Incarcerated individuals.
13. Non-English speaking subjects.
14. Participant's weight must be </= 350 lbs.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Participant-Reported Safety and Efficacy Following Use of Investigational Device | From device use through completion of the final study visit, up to one year
  The number of participants who report any device-related safety concerns following use of the investigational non-significant risk device, as assessed by participant-reported surveys.

SECONDARY OUTCOMES:
Participants with Osteoarthritic Joints Reaction to the LFU | one year
  To determine the potential impact the device may have on patients as their osteoarthritic joints react to the LFU, which will be denoted by surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blackwell, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States